CLINICAL TRIAL: NCT05568160
Title: Prospective Randomized Double-blind Study Evaluating the Superiority of VAsopressin Versus NOradrenaline in the Management of Patients at Risk of Kidney Failure Undergoing Cardiac Surgery With Extracorporeal Circulation
Brief Title: Evaluation of the Superiority of VAsopressin Versus NOradrenaline in the Management of Patients at Risk of Kidney Failure Undergoing Cardiac Surgery With Extracorporeal Circulation
Acronym: NOVACC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GUINOT PHRCI 2019
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Scheduled Cardiac Surgery With Extracorporeal Circulation; Vasoplegic Syndrome
MeSH Terms: conditions — Vasoplegia | interventions — Vasopressins; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Drug: Vasopressin; Other: Collection of clinical data; Other: Quality of Life Questionnaire EQ-5D
- Control (Active Comparator)
  Interventions: Drug: Norepinephrine; Other: Collection of clinical data; Other: Quality of Life Questionnaire EQ-5D

INTERVENTIONS:
Drug: Vasopressin — The infusion is started at 5 ml hr-1, increased in increments of 1 ml hr-1 every 5 minutes to reach a maximum target rate of 30 ml hr-1
  Arms: Intervention
Drug: Norepinephrine — The infusion is started at 5 ml h-1, increased in increments of 1 ml h-1 every 5 minutes to a maximum target rate of 30 ml h-1
  Arms: Control
Other: Collection of clinical data — At D1, D2, D7, D30 or D60 and D90
Other: Quality of Life Questionnaire EQ-5D — At the anesthesia consultation, discharge from intensive care, D7, D30 and D90

SUMMARY:
This is a randomized, double blind, multicenter study following surgery with extracorporeal circulation to compare blood pressure optimization with vasopressin versus noradrenaline. It is planned to include 840 patients in order to have 420 patients with vasoplegic syndrome.

The primary objective of this study is to determine whether the use of vasopressin to maintain blood pressure following cardiac surgery decreases the number of patients with acute renal failure and/or death compared with the usual use of norepinephrine.

Participation in the study involves daily follow-up at D1, D2, and D7 of the onset of the syndrome and then follow-up at D30 and D90.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has given free, written and informed consent
* Patient of legal age.
* Negative pregnancy test for women of childbearing age
* Patient requiring cardiac surgery:

  * Scheduled (> 24h)
  * With extracorporeal circulation (ECC)
  * Myocardial revascularization (coronary bypass), and/or surgical correction of valvulopathy (aortic, mitral, pulmonary, tricupsidian), and/or of the ascending aorta and/or removal of an intracardiac tumor, and/or closure of a PFO/ASD
* Patient with at least 3 risk factors for acute kidney failure including:

  * age > 70 years, combined surgery (more than two procedures), common trunk lesion, preoperative anemia, chronic respiratory failure, obliterative arterial disease of the lower extremities, diabetes, glomerular filtration < 60 ml min-1 m², LVEF <40%, redux, intra-aortic counterpulsation balloon, expected duration of bypass surgery > 100 min, albuminuria

Exclusion Criteria:

* Patient not affiliated to national health insurance or not beneficiary of a social security system,
* Patient subject to a measure of legal protection (curatorship, guardianship),
* Pregnant, parturient or breastfeeding women,
* Patients of legal age who are incapable or unable to express their consent,
* Patients who have already been included in this study
* Patients requiring emergency surgery (less than 24 hours)
* Patient with chronic kidney failure on dialysis,
* Patient with a cardiac transplant,
* Patient on left-sided monoventricular assistance,
* Patient on ECMO/ECLS,
* Patient with acute circulatory failure in the immediate preoperative period (sepsis, hemorrhage),
* Patients with known hypersensitivity to the active ingredient (argipressin) or to one of the excipients of REVERPLEG®.

Secondary exclusion criteria:

* Patient not developing persistent arterial hypotension (vasoplegic syndrome), within 12 hours after completion of surgery, defined as persistent mean arterial pressure (MAP) <65 mmHg despite correction of preload and inotropism, with a cardiac index >2.2 l min-1 m-2, and not responding to 30 mg cumulative of ephedrine in bolus
* Patient with hemorrhagic shock perioperatively before receiving vasopressor therapy (treatment under study)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a renal complication or death | From the onset of the vasoplegic syndrome until 7 days after

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Derived] Guinot PG, Desebbe O, Besch G, Guerci P, Gaudard P, Lena D, Mertes PM, Abou-Arab O, Bouhemad B; NOVACC study group. Prospective randomized double-blind study to evaluate the superiority of Vasopressin versus Norepinephrine in the management of the patient at renal risk undergoing cardiac surgery with cardiopulmonary bypass (NOVACC trial). Am Heart J. 2024 Jun;272:86-95. doi: 10.1016/j.ahj.2024.03.008. Epub 2024 Mar 16. PMID 38492626